CLINICAL TRIAL: NCT01207531
Title: miRNA in the Evaluation of the Value of Sepsis Prognosis Prospective Observational Study
Brief Title: MiRNAs Evaluate the Prognosis of Sepsis
Acronym: METPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Pneumology Department of Chinese PLA General Hospital
Other Study IDs: 301PLAGH-2010915
Record Dates: First submitted 2010-09-17; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Sepsis
Keywords: sepsis; miRNA
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Survival Group
- Death group

SUMMARY:
Sepsis is a common cause of death in intensive care unit, timely and accurate diagnosis and treatment directly affect the survival rate. MiRNA is a post-transcriptional small RNA which regulate mRNA expression. The present study was designed to screen several miRNA by microarray which evaluate the sepsis prognosis in order to be a new target for the treatment of sepsis.

DETAILED DESCRIPTION:
The study is a non-intervention, prospective observational study. Purpose of this sudy is to screening several miRNAs by microarray which can evaluate the prognosis of sepsis . We will collect serum samples from patients with sepsis in SICU, RICU and EICU of 301 Hospital since September 2009 , and then use the chip and qRT-PCR to Screen miRNAs which can evaluate the prognosis of sepsis, and statistical analysis the miRNAS expression correlation with SOFA score.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sepsis
* Patients who agree with the study

Exclusion Criteria:

* Aged <18 years;
* Into the group who died within 24 hours;
* Agranulocytosis (<0.5 × 109 / L);
* Combined HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: within 24 hours after admited in ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-11 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 28days after admited in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, Doctor, Study Director — Pneumology Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang H, Zhang P, Chen W, Feng D, Jia Y, Xie L. Serum microRNA signatures identified by Solexa sequencing predict sepsis patients' mortality: a prospective observational study. PLoS One. 2012;7(6):e38885. doi: 10.1371/journal.pone.0038885. Epub 2012 Jun 15. PMID 22719975